CLINICAL TRIAL: NCT00895544
Title: An Open-Label Phase 1/2 Study to Assess the Immunogenicity and Safety of a Single Prime-Boost Vaccination Schedule With a Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine in Healthy Volunteers Aged 18 to 59 Years
Brief Title: Immunogenicity and Safety Study of a Single Prime-Boost Vaccination Schedule With a H5N1 Influenza Vaccine in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Gerald Aichinger, MD; Study Medical Director, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 810802
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2011-07

CONDITIONS: Influenza; Avian Influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Day 0: Single priming vaccination with Dose A of whole virion, Vero cell-derived influenza vaccine (Vietnam strain) - Day 360: Randomization to booster vaccination with Dose B of whole virion, Vero cell-derived influenza vaccine (Indonesia strain)
  Interventions: Biological: Influenza vaccine (whole virion, Vero cell derived)
- 2 (Experimental): Day 0: Single priming vaccination with Dose A of whole virion, Vero cell-derived influenza vaccine (Vietnam strain) - Day 360: Randomization to booster vaccination with Dose A of whole virion, Vero cell-derived influenza vaccine (Indonesia strain)
  Interventions: Biological: Influenza vaccine (whole virion, Vero cell derived)

INTERVENTIONS:
Biological: Influenza vaccine (whole virion, Vero cell derived) — Dose A (Vietnam strain) for priming vaccination (Day 0) - Dose B (Indonesia strain) for booster vaccination (Day 360)
  Arms: 1
Biological: Influenza vaccine (whole virion, Vero cell derived) — Dose A (Vietnam strain) for priming vaccination (Day 0) - Dose A (Indonesia strain) for booster vaccination (Day 360)
  Arms: 2

SUMMARY:
The main objective of the study is to assess the immune response to a non-adjuvanted H5N1 influenza vaccine in an adult population when administered according to a single prime-boost schedule.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if they:

* are 18 to 59 years of age, inclusive, on the day of screening
* have an understanding of the study and its procedures, agree to its provisions, and give written informed consent prior to study entry
* are generally healthy, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination
* are physically and mentally capable of participating in the study and follow its procedures
* agree to keep a daily record of symptoms for the duration of the study
* if female of childbearing potential: have a negative urine pregnancy test result within 24 hours prior to the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* have a history of exposure to H5N1 virus or a history of vaccination with an H5N1 influenza vaccine
* are at high risk of contracting H5N1 influenza infection (e.g. poultry workers)
* currently have or have a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* have any inherited or acquired immunodeficiency
* have a disease or are currently undergoing a form of treatment or were undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (> 800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* have a history of severe allergic reactions or anaphylaxis
* have a rash, dermatological condition or tattoos which may interfere with injection site reaction rating
* have received any blood products or immunoglobulins within 90 days prior to study entry
* have donated blood or plasma within 30 days prior to study entry
* have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study
* have a functional or surgical asplenia
* have a known or suspected problem with alcohol or drug abuse
* were administered an investigational drug within 6 weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* are a member of the team conducting this study or are in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study
* if female: are pregnant or lactating

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain associated with protection 21 days after the booster vaccination defined as titer measured by microneutralization test >= 1:20. | 21 days

SECONDARY OUTCOMES:
Number of subjects with antibody response associated with protection 21, 42, 180 and 360 days after the priming vaccination and 21 days after the booster vaccination | at the timepoints stated above

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Aichinger, MD, Study Director — Baxter Healthcare Corporation
Locations (3):
- General Hospital of Vienna (AKH Wien), Dept. of Clinical Pharmacology, Vienna, Austria
- Finland (2):
  - Espoon rokotetutkumusklinikka, Espoo
  - Etelä - Helsingin rokotetutkimusklinikka, Helsinki